CLINICAL TRIAL: NCT01515202
Title: A Randomized, Placebo-Controlled, Double-Blinded, Multiple Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-823778 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: Japanese Phase 1 Multiple Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB121-009
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BMS-823778

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Panel 1: BMS-823778 or Placebo matching BMS-823778 (Experimental): Healthy Subjects
  Interventions: Drug: BMS-823778; Drug: Placebo matching with BMS-823778
- Panel 2: BMS-823778 or Placebo matching BMS-823778 (Experimental): Healthy Subjects
  Interventions: Drug: BMS-823778; Drug: Placebo matching with BMS-823778
- Panel 3: BMS-823778 or Placebo matching BMS-823778 (Experimental): Healthy Subjects
  Interventions: Drug: BMS-823778; Drug: Placebo matching with BMS-823778
- Panel 4: BMS-823778 or Placebo matching BMS-823778 (Experimental): Subjects with T2DM
  Interventions: Drug: BMS-823778; Drug: Placebo matching with BMS-823778
- Panel 5: BMS-823778 or Placebo matching BMS-823778 (Experimental): Subjects with T2DM
  Interventions: Drug: BMS-823778; Drug: Placebo matching with BMS-823778

INTERVENTIONS:
Drug: BMS-823778 — Capsules, Oral, 2 mg, Once daily, 14 days
  Arms: Panel 1: BMS-823778 or Placebo matching BMS-823778; Panel 4: BMS-823778 or Placebo matching BMS-823778
Drug: BMS-823778 — Capsules, Oral, 12 mg, Once daily, 14 days
  Arms: Panel 2: BMS-823778 or Placebo matching BMS-823778
Drug: BMS-823778 — Capsules, Oral, 25 mg, Once daily, 14 days
  Arms: Panel 3: BMS-823778 or Placebo matching BMS-823778
Drug: BMS-823778 — Capsules, Oral, 15 mg, Once daily, 14 days
  Arms: Panel 5: BMS-823778 or Placebo matching BMS-823778
Drug: Placebo matching with BMS-823778 — Capsules, Oral, 0 mg, Once daily, 14 days

SUMMARY:
The purpose of this clinical study is to assess the safety and tolerability of multiple oral doses of BMS-823778 in healthy Japanese subjects and Japanese patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
MAD study - Multiple Ascending Dose study

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with Type 2 Diabetes Mellitus (T2DM) [Fasting glucose < 240 mg/dL, Hemoglobin A1c (HbA1c): 6.5% to 10.0% National Glycohemoglobin Standardization Program (NGSP)] who are treatment-naive and managed with diet and/or exercises only, ages: 20 to 65 years

Exclusion Criteria:

* Patient who is taking any medication for T2DM
* Symptoms of poorly controlled diabetes that would preclude participation in this placebo-controlled trial
* Insulin therapy within one year of screening

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by the number, frequency and intensity of adverse events, vital sign measurements, ECGs, physical examinations, and clinical laboratory tests | Up to Day 21

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Trough observed plasma concentration (Cmin) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Time of maximum observed plasma concentration (Tmax) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Area under the plasma concentration-time curve in one dosing interval [AUC(TAU)] of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Accumulation Index following multiple dosing (AI) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Plasma half-life (T-HALF) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Percent urinary recovery (% UR) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Apparent total body clearance (CLT/F) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Renal clearance from plasma (CLR) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Peak to trough ratio (Cmax/Cmin) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Effective plasma half-life (T-HALFeff) of BMS-823778, as measured by plasma/urine concentration | Up to Day 21
Pharmacodynamics, as measured by Serum concentration of cortisol and cortisone after an oral dose of cortisone and biomarkers for HPA axis activity (urinary free cortisol and cortisone, salivary cortisol, ACTH, DHEA-S and 4-androstenedione) | Up to Day 21
  * HPA = Hypothalamic-pituitary-adrenal
  * DHEA-S = Dehydroepiandrosterone-sulphate
  * ACTH = adrenocorticotropic hormone

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Hachioji-Shi, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx